CLINICAL TRIAL: NCT00005567
Title: Parental Knowledge and Beliefs About Infant Sleep Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Educational/Counseling/Training
Other Study IDs: NCRR-M01RR06022-0038; M01RR006022 (NIH)
Record Dates: First submitted 2000-04-22; First posted 2000-04-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: Sudden Infant Death Syndrome
MeSH Terms: conditions — Sudden Infant Death

INTERVENTIONS:
Behavioral: Parental knowledge and beliefs about infant sleep position

SUMMARY:
In the United States, Sudden Infant Death Syndrome (SIDS)is the leading cause of death in infants between the ages of 1 and 12 months. The etiology of SIDS is still not clear although a number of risk factors have been identified. Sleeping on the stomach has been identified as a major risk for SIDS. The rates of SIDS have dropped substantially in countries in which the usual sleep position has changed from the stomach to the side or back. Back sleep has been shown to be the most stable and safest position. The American Academy of Pediatrics now recommends the back sleeping position for all healthy infants. Since the American Academy of Pediatrics began advocating the back sleep position, the incidence of SIDS has decreased by more than 40% in this country. However, the decrease has not been uniform across segments of the population. Black infants continue to have a higher rate of SIDS compared with other groups. This discrepancy could be related to infant sleep position practices. Several studies have shown that infants born to low income, minority, inner-city families were more likely to be placed on the stomach to sleep. Education appears to influence choice of sleep position and may explain, at least to some degree, the difference in choice of sleep position among certain groups. We believe that uniform education of parents will influence the sleep position that parents choose for their baby. We will undertake this initial study to document what parents choose to do with their infants regarding sleep position and why they make these choices so that we can improve our educational approach.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a two-week old infant born in the Well Newborn Nursery at Yale-New Haven Hospital. Infant is brought for well child care at Yale-New Haven Hospital Primary Care Center

Ages: 0 Years to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child